CLINICAL TRIAL: NCT02422355
Title: A Focused Registry on the Femoral Neck System (FNS) in Patients With Femoral Neck Fractures
Acronym: FR_FNS
Status: Completed | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: FR FNS
Record Dates: First submitted 2015-03-27; First posted 2015-04-21 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2021-12

CONDITIONS: Femoral Neck Fracture; Hip Fracture
Keywords: hip; femoral neck; Garden classification; healing; cut-out; iatrogenic fracture; implant; rotational stability; minimal invasive
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Femoral Neck Fractures AO/OTA 31-B1:3: Fixation using the implant FNS.
  Interventions: Device: FNS

INTERVENTIONS:
Device: FNS — Surgical intervention using the FNS

SUMMARY:
In comparison to previous implants, the Femoral neck system (FNS) is an approved implant by the competent authorities (CE mark). It is designated to stabilize medial femoral neck fractures in a minimal invasive technique. The implant combines an angular stable device with screw in screw technology for rotational stability. Therefore the purpose of this focused registry is to investigate how the newly developed and approved implant called FNS is performing clinically and radiologically in terms of surgical technique, intra- and postoperative complications and short term outcome.

DETAILED DESCRIPTION:
All patients included are treated as per standard or care and followed up from the time point of enrollment until at least three months after surgery as described below. Data of a visit after 6 months and 12 months are collected if bone union according to the RUSH score is not complete after 3 or 6 months respectively or if the patient has persistent or increasing pain on the operated site.

Preoperative:

* Patient details
* Fracture Classification and comminution based on CT
* Pre-fracture HHS and EQ5D
* X-rays

Intraoperative:

* Surgery details
* Defined intraoperative complications
* Intraoperative fluoroscopy: hip ap (with leg 15° internally rotated) and lateral after reduction and after implant placement

Postoperative:

* X-ray prior to any mechanical load: hip ap (with leg 15° internally rotated) and lateral

  6 weeks and 3 months FU:
* Defined postoperative complications
* HSS and EQ5D
* X-rays

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of a medial femoral neck fracture (AO/OTA 31-B1:3) with the need of a fixation using the FNS.
* Ability to understand the content of the patient information/Informed Consent Form
* Willingness and ability to participate in the registry according to the Registry Plan (RP)
* Signed and dated Ethics Committee (EC)/Institutional Review Board (IRB) approved written informed consent

Exclusion Criteria:

* Pathological fracture
* Additional acute fracture
* Any not medically managed severe systemic disease
* Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the registry period
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from a femoral neck fracture (AO/OTA 31-B1:3) with the need of a fixation using the FNS.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of complications within the first 3 months after surgery | 3 months

SECONDARY OUTCOMES:
Fracture mechanism | Pre-operatively (Day -1)
  Classification of the fracture mechanism in one of the following group: Fall from standing height , Falls from elevated height, Road traffic accident or Other causes
Classification of the fracture | Pre-operatively (Day -1)
  Classification of the fracture using the Garden classification and the AO/AOTA classification
Time from injury to surgery | Surgery (Day 0)
  Time in hours from the injury to the start of the surgery
Length of surgery | Surgery (Day 0)
  Time in minutes from first incision to closure
Harris Hip Score | Pre-operatively (Day -1), 6 weeks, 3 months, 6 months and 12 months after surgery
EQ5D-5L | Pre-operatively (Day -1), 6 weeks, 3 months, 6 months and 12 months after surgery
Radiological bone union (RUSH score) | 6 weeks, 3 months, 6 months and 12 months after surgery
  RUSH score
Quality of reduction (Garden's alignment index and Lowell's criteria) | Surgery (Day 0)
  Garden's alignment index and Lowell's criteria

CONTACTS AND LOCATIONS:
Overall Officials: Karl Stoffel, Prof, Principal Investigator — Cantonal Hosptal, Baselland
Locations (7):
- Medizinische Universität Innsbruck, Innsbruck, Tyrol, Austria
- Germany (2):
  - Ulm University, Ulm, Baden-Wurttemberg
  - Friedrich-Schiller-Universität Jena, Jena, Thuringia
- Switzerland (4):
  - Kantonsspital Baselland, Bruderholz, Basel-Landschaft
  - Ospedale Regionale di Lugano, Lugano, Canton Ticino
  - Luzerner Kantonsspital, Lucerne
  - Stadtspital Triemli, Zurich

REFERENCES:
- [Derived] Stoffel K, Michelitsch C, Arora R, Babst R, Candrian C, Eickhoff A, Gebhard F, Platz A, Schmid FA, Weschenfelder W, Sommer C. Clinical performance of the Femoral Neck System within 1 year in 125 patients with acute femoral neck fractures, a prospective observational case series. Arch Orthop Trauma Surg. 2023 Jul;143(7):4155-4164. doi: 10.1007/s00402-022-04686-w. Epub 2022 Dec 2. PMID 36460761
- See also: Sponsor's website — https://www.aofoundation.org